CLINICAL TRIAL: NCT07200349
Title: Clinical Evaluation of Local Calcitriol Delivery on Maxillary Canine Retraction
Acronym: CALCR25
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Taha Ahmed Hassan, Postgraduate Researcher (Master's Candidate), Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZH2025CalcitriolCR
Record Dates: First submitted 2025-07-30; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-07

CONDITIONS: Maxillary Canine Retraction; Local Calcitriol Delivery; Orthodontic Tooth Movement
Keywords: Calcitriol; Vitamin D3; Canine Retraction; Split-mouth Trial

STUDY DESIGN:
Intervention Model Description: This is a parallel design with two groups based on Vitamin D status. Each participant receives a split-mouth intervention with Calcitriol on one side and no treatment on the other side
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D Sufficient Group (Experimental): Patients with normal serum vitamin D levels. Each patient receives a local Calcitriol delivery on one side of the maxilla, and the other side serves as control (split-mouth).
  Interventions: Drug: Calcitriol Delivery
- Vitamin D Deficient Group (Experimental): Patients with normal serum vitamin D levels. Each patient receives a local Calcitriol delivery on one side of the maxilla, and the other side serves as control (split-mouth).
  Interventions: Drug: Calcitriol Delivery

INTERVENTIONS:
Drug: Calcitriol Delivery — Local delivery of Calcitriol (active form of vitamin D3) to one side of the maxillary canine area during orthodontic treatment. The aim is to assess its effect on dental and skeletal changes during canine retraction in a split-mouth design.

SUMMARY:
This study will evaluate the effect of locally applied Calcitriol on dental and skeletal changes during upper canine retraction. It is a split-mouth randomized clinical trial, where Calcitriol will be locally applied on one side of the maxilla, and the other side will serve as control.

DETAILED DESCRIPTION:
Orthodontic tooth movement depends on bone remodeling. This study investigates if Calcitriol, the active form of vitamin D3, can affect this process when applied locally during upper canine retraction. The study is designed as a split-mouth randomized clinical trial. Patients needing maxillary first premolar extraction will be included. Calcitriol will be locally applied on one side, and the other will serve as a control. The study will evaluate dental and skeletal changes to see if Calcitriol improves treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of class I malocclusion requiring bilateral extraction of the maxillary first premolars and subsequent canine retraction.
2. Presence of class II malocclusion requiring bilateral extraction of the maxillary first premolars and subsequent canine retraction.
3. Age range between 13 and 35 years to include both adolescent and adult patients suitable for orthodontic treatment.
4. Presence of permanent dentition.
5. Good oral hygiene.

Exclusion Criteria:

1. History of chronic systemic disease.
2. Presence of active gingival or periodontal disease.
3. Known allergy or hypersensitivity to vitamin D.
4. Pregnancy or lactation.
5. History of previous orthodontic treatment.
6. Presence of craniofacial anomalies affecting bone physiology.

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Amount of maxillary canine retraction (mm) assessed on CBCT scans | T0: immediately before maxillary canine retraction. T1: after completion of canine retraction (approximately 4 months - 6 months)
  The amount of maxillary canine movement will be assessed using cone-beam computed tomography (CBCT). Measurements will be expressed in millimeters

IPD SHARING:
Plan to Share IPD: No
This is a university-based academic study conducted as part of a master's thesis. There is no plan to share individual participant data due to the absence of a data-sharing agreement or external funding